CLINICAL TRIAL: NCT01895738
Title: WrapAround Care for Youth Injured by Violence: A Pilot Randomized Control Trial
Brief Title: WrapAround Care for Youth Injured by Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Carolyn Snider, Assistant Professor, Department of Emergency Medicine, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H2013:257; 302030 (Other Grant/Funding Number: Canadian Institute of Health Research)
Record Dates: First submitted 2013-07-04; First posted 2013-07-10 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Trauma; Injuries; Violence
Keywords: Trauma; Injuries; Violence; Adolescent; WrapAround care
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WrapAround Care (Experimental): Participants randomized to the intervention arm will be met in the emergency department by a support worker who has lived experience. They will start to build a relationship with the participant at that time (i.e. during the teachable moment) and will work with the participant for approximately one year, delivering WrapAround Care. Wraparound care is an established care model that starts with linking an individual with a support￼￼￼ worker who works with them to address risk factors and enable the individual to make positive choices. It is hypothesized that by working with youth to address the risk factors in their control, the likelihood of future violence is reduced.
  Interventions: Behavioral: WrapAround Care
- Standard of Care (No Intervention): Standard of Care is typically a sheet of community resources potentially handed out by the emergency physician, nurse or social worker.

INTERVENTIONS:
Behavioral: WrapAround Care — Wraparound care is an established care model that starts with linking an individual with a support￼￼￼ worker who works with them to address risk factors and enable the individual to make positive choices. It is hypothesized that by working with youth to address the risk factors in their control, the likelihood of future violence is reduced.
  Arms: WrapAround Care

SUMMARY:
Youth injured by violence is a major public health concern in Canada. It is the fourth cause of death and the leading reason for a youth to visit an emergency department (ED). In Winnipeg, 20% of youth who visit an emergency department with an injury due to violence have a second visit for a subsequent violent injury within the following year. This is consistent with studies in other jurisdictions that demonstrate that violent injury is a chronic condition. Youth injured by violence are in a reflective and receptive state of mind, rendering the emergency department setting appropriate for intervention. The investigators propose a WrapAround Care model delivered by a support worker with lived experience with violence, supported by a social worker, an addictions and mental health counsellor, a family counsellor and links to multiple community partners. Support workers will be on call 24 hours a day, 7 days a week in order to start the intervention in the ED and take advantage of the "teachable moment". The proposed study is a pilot randomized control trial to assess the feasibility of a randomized control trial designed to assess efficacy. For the pilot trial the investigators will assess recruitment, treatment fidelity, participant adherence and safety. The intervention arm will receive wraparound care initiated at the time of their visit for injury due to violence. The control arm will receive standard of care (usually a list of community contacts). The investigators will use an adapted pre-consent randomization methodology. This intervention has been developed using a community based participatory research approach. Our team includes clinicians, nurses, social workers, community youth workers, ex-gang members, elders and researchers.

DETAILED DESCRIPTION:
Youth injured by violence is a major public health concern in Canada. It is the fourth cause of death and the leading reason for a youth to visit an emergency department. In Winnipeg 20% of youth who visit an emergency department with an injury due to violence have a second visit for a subsequent violent injury within the following year. This is consistent with studies in other jurisdictions that demonstrated that violent injury is a chronic condition.

Youth injured by violence have been shown to be in a reflective and receptive state of mind, rendering the emergency department setting appropriate for intervention. There are some hospital-based intervention programs for youth injured by violence in the U.S.; however, they have not been evaluated to assess repeat injury using a randomized control trial (RCT) and given the cost of this intervention, significant equipoise exists. It is essential to evaluate this intervention rigorously using RCT methodology. A pilot RCT is prudent prior to the main RCT.

The investigators propose a WrapAround Care model delivered by a support worker with lived experience with violence, supported by a social worker, an addictions and mental health counsellor, a family counsellor and links to multiple community supports. These community supports include partnerships with aboriginal and newcomer youth cultural programs as many youth impacted by violence are aboriginal and new immigrants to Canada. Support workers will be on call 24 hours a day, 7 days a week in order to start the intervention in the ED and take advantage of the "teachable moment".

This pilot study RCT will enroll 180 youth (aged 14 - 24) over one year (90 to each arm). The treatment arm will be the WrapAround care model initiated at the time of injury (i.e. in the emergency department). The control arm will be providing youth with a list of community programs and will be a waitlist control. The primary outcomes of the pilot study will evaluate evaluate recruitment, adherence, fidelity and safety of the intervention. The primary outcome for the main trial is repeat visit to any emergency department in Winnipeg for a subsequent injury due to interpersonal violence. This will be measured using a combination of administrative data and chart review to ensure high follow-up. The secondary outcomes include measurement of counts and severity of injury and housing and education changes. This intervention has been developed using a community based participatory research approach. Our team includes clinicians, nurses, social workers, community youth workers, former gang members, elders and researchers.

ELIGIBILITY:
Inclusion Criteria:

* Age 14 - 24 AND
* Presentation with an injury caused by violence (defined as an injury inflicted by someone else and one of a gunshot wound, stab wound, injury due to blunt object, or injury due to bodily force)

Exclusion Criteria:

* Unable to consent due to language or brain injury
* Sexual assault (except those explicitly described as gang related - being "raped in or raped out" of a gang which is common with female gang members)
* Child Abuse
* Self-Inflicted Injury
* Transfer from a hospital > 1 hour from Winnipeg.

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 133 (Actual)
Dates: Start 2013-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of Recruitment for Main Trial | One Year
  The investigators estimate that our sample size for the main trial must be 330 per arm (660 total) (Section 2.11). In order to ensure sufficient recruitment over 44 months plus 12 month follow-up for each subject and analysis time within a 5 year time frame, the investigators estimate that the investigators will need to randomize 180 youth to our pilot study in one year. This will also ensure that each support worker has an appropriate workload (approximately 2 new subjects per month with a maximum of 15 at any time). Successful Recruitment will be defined as >180 participants in one year.
Fidelity to Treatment Protocol | Two Years
  The investigators have set the treatment protocol based on experience from our Proof of Concept study and our community partners. In behavioural interventions, fidelity measures are considered the quality control measure of ensuring the intervention is being implemented as intended. Fidelity preserves internal validity against type I and II errors, it improves power by decreasing the variability in treatment effect and allows replication, dissemination and implementation in practice. Successful Fidelity will be defined as >85% of contacts (i.e. check-ins, phone calls, team meetings) attempted by the support worker.
Participant Adherence | Two Years
  Participant adherence refers to both the receipt of the intervention (the development of a strong and effective alliance between the case manager and youth) and enacting on the intervention (accessing resources). In behavioural intervention studies it is important to demonstrate that the actual intervention is occurring as designed. If adherence to the intervention is not achieved, then our comparison of outcomes do not truly measure the difference between intervention and control. Successful Adherence will be assessed using the Working Alliance Inventory, which measures the bond between the support worker and participant and the agreement on tasks and goals set.
Serious Adverse Events | Two Years
  Given youth injured by violence, especially those who are gang-involved are at high risk of retaliatory violence; investigators must ensure participants do not experience increased harm as part of the intervention. Program staff will discuss adverse events at each weekly meeting and workers and counselors will be required to fill in adverse event forms should they occur. These will be reviewed immediately with the principal investigator and if necessary the Data Safety Monitoring Board (DSMB). The DSMB will review a table of these adverse events and will review serious adverse events (e.g. death or otherwise deemed as serious) in detail. Stopping rules and guidelines are specified for the DSMB. The main stopping rule will be to stop the study if the treatment arm is significantly more likely to suffer a repeat violent injury (p<0.05).

SECONDARY OUTCOMES:
To determine the cost-effectiveness of the intervention | Two Years
  This outcome is designed to determine the cost-effectiveness of this intervention. For this pilot study we will only be including the direct costs of repeat visits to the hospital for injury, substance use and mental health. The purpose of this initial assessment is to support future cost-effectiveness study of our main study.

OTHER OUTCOMES:
To determine the impact on Visits to Hospital for Repeat Intentional Injury within one year | Two Years
  This will be the primary outcome for our future effectiveness trial - we will measure this in our pilot trial to ensure data is collectible and appropriate for analysis
  20% of youth who visit the Winnipeg Health Science EDs for a visit due to violence have a subsequent visit to the same ED for a new injury due to violence in the following year. This is similar to figures from other locations in North America and Europe, which have demonstrated repeat injury rates as high as 40%.
To determine the impact on # of repeat intentional injuries | Two Years
  This will be a secondary outcome of our future effectiveness trials - we will measure this in our pilot trial to ensure data is collectible and appropriate for analysis.
  Of the youth who had subsequent visits to our EDs for injuries due to violence, 81% had >1 repeat injury and 21% had >2 repeat injuries.8 This outcome will determine if the intervention has an impact on number of repeat intentional injuries.
To determine the impact on time to repeat intentional injury | Two Years
  This will be a secondary outcome of our future effectiveness trials - we will measure this in our pilot trial to ensure data is collectible and appropriate for analysis
  One study demonstrated that a person is at highest risk of reinjury in the first 30 days. This outcome will determine if the intervention protects from early repeat reinjury.
To determine the impact on severity of repeat injury | Two Years
  This will be a secondary outcome of our future effectiveness trials - we will measure this in our pilot trial to ensure data is collectible and appropriate for analysis
  It is hypothesized that subsequent injuries are more severe; however, no literature exists to prove this hypothesis. We will use the Injury Severity Score and the Abbreviated Injury Scale to measure this. This outcome will determine if the intervention protects from more serious repeat injury.
To determine the impact on visits to hospital related to substance use | Two Years
  This will be a secondary outcome of our future effectiveness trials - we will measure this in our pilot trial to ensure data is collectible and appropriate for analysis.
To determine the impact on visits to hospital for mental health care | Two Years
  This will be a secondary outcome of our future effectiveness trials - we will measure this in our pilot trial to ensure data is collectible and appropriate for analysis
To determine the impact on education | Two Years
  This will be a secondary outcome of our future effectiveness trials - we will measure this in our pilot trial to ensure data is collectible and appropriate for analysis
  Education is associated with reduced violence involvement. We will measure whether the youth was enrolled in either high school or post-secondary education at both time of index injury and at the end of one year. This outcome will determine if the intervention is successful in addressing this risk factor.
To determine the impact on housing | Two Years
  This will be a secondary outcome of our future effectiveness trials - we will measure this in our pilot trial to ensure data is collectible and appropriate for analysis
  Many injured faced a lack of stable housing. This means that the youth is often "couch surfing" or staying in dangerous environments or on the street. We will measure whether the youth was housed in public housing at both time of index injury and at the end of one year.
To determine the impact on criminal behaviour | Two Years
  This will be a secondary outcome of our future effectiveness trials - we will measure this in our pilot trial to ensure data is collectible and appropriate for analysis
  Previous incarceration has been associated with increased risk of violent injury and homicide. Other literature demonstrates that violent injury in youth may precede criminal behaviour. We will measure interactions with the Manitoba Justice system in the year prior to the index injury and the year post the index injury to determine if the intervention protects the youth from interactions with Manitoba Justice.
To determine the impact on repeat injuries due to violence by self-report | Two Years
  This will be a secondary outcome of our future effectiveness trials - we will measure this in our pilot trial to ensure data is collectible and appropriate for analysis
  Some repeat injuries that occur will not be severe enough to require a visit to an ED; youth may visit their family physician, a walk-in-clinic or not require any medical care. We will measure injuries not captured by hospital administrative data and chart review by asking youth to self-report these injuries to determine if the intervention causes changes in self-report of repeat injury.
To determine the impact on structured activity by self-report | Two Years
  This will be a secondary outcome of our future effectiveness trials - we will measure this in our pilot trial to ensure data is collectible and appropriate for analysis
  Structured activity - as defined as being in school, in job training, employed or volunteering is important to helping youth be more future oriented. We will measure this each month to determine if the intervention causes changes in self-report of structured activity.
To determine the impact on housing by self-report | Two Years
  This will be a secondary outcome of our future effectiveness trials - we will measure this in our pilot trial to ensure data is collectible and appropriate for analysis
  As noted in previous secondary outcomes, safe housing is challenging for our participants. Some may find safe housing through private landlords and therefore not be measured in the administrative database. We will measure their self-report of being safely housed to determine if the intervention promotes safe housing.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Snider, MD MPH, Principal Investigator — University of Manitoba
Locations (1):
- Winnipeg Health Sciences Centre, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Snider C, Jiang D, Logsetty S, Strome T, Klassen T. Wraparound care for youth injured by violence: study protocol for a pilot randomised control trial. BMJ Open. 2015 May 19;5(5):e008088. doi: 10.1136/bmjopen-2015-008088. PMID 25991461